CLINICAL TRIAL: NCT06546644
Title: Effect of a Structured School-based Health Intervention for Obesity Prevention In Children Aged 5-12 Years
Brief Title: A Structured School-based Health Intervention for the Obesity Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FAHS
Record Dates: First submitted 2024-08-03; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Child Obesity; Child Behavior; Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity; Child Behavior

STUDY DESIGN:
Intervention Model Description: The participants after baseline measures, will be randomly assigned into two groups intervention and control in a parallel way.
Who Masked: Outcomes Assessor
Masking Description: Only the Outcomes Assessor will be blinded regarding group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The children in the intervention group will receive a school-based structured health intervention to prevent obesity in children aged 5-12 years. A pre-tested validated structured school-based intervention is developed for children in the intervention group. The intervention included behavior change regarding dietary patterns and physical activity. Education will be provided to children in lectures, PowerPoint, smart handouts, and videos. The parents will also be involved in this educational stream through seminars and parent schools specially organized events.
  Interventions: Behavioral: Structured school-based intervention
- Control (No Intervention): The children in the control group will receive no intervention.

INTERVENTIONS:
Behavioral: Structured school-based intervention — A pre-tested validated structured school-based intervention is developed for children in the intervention group. The intervention included behavior change regarding dietary patterns and physical activity. Education will be provided to children in lectures, PowerPoint, smart handouts, and videos. The parents will also be involved in this educational stream through seminars and parent schools specially organized events.
  Arms: Intervention group

SUMMARY:
The proposed research aims to assess how well a structured intervention is intended to reduce childhood obesity. The intervention addresses food and physical activity behaviors, important determinants of obesity, by concentrating on these elements. The goal of nutritional and physical education is to raise knowledge about the negative effects of obesity and encourage healthy eating habits in children and their caregivers. These educational campaigns will be delivered primarily through schools, guaranteeing a wide audience and consistent messaging.

DETAILED DESCRIPTION:
The demographic profile of Pakistan offers a unique background for researching the dynamics of childhood obesity because of its rapid urban growth and socioeconomic shifts. Processed foods are displacing traditional diets, and children's physical activity is decreasing as a result of longer screen times and restricted access to leisure centers.

The proposed research aims to assess how well a structured intervention is intended to reduce childhood obesity. The intervention addresses food and physical activity behaviors, important determinants of obesity, by concentrating on these elements. Dietary Education: Teaches kids about eating the right portions of food and maintaining a balanced diet. Better eating habits and an understanding of nutrition are among the results.

Information regarding Physical Activity: Raises awareness and encourages regular exercise. Improved comprehension and engagement in physical activities are among the results.

Extra Physical Activity Time: Offers extra opportunities for physical activity after school, such as fitness classes and sports, after hours. Improved fitness, a decrease in sedentary time, and higher levels of physical activity are the results.

ELIGIBILITY:
Inclusion Criteria:

* Children of age between 5 to 12 years.
* Enrollment at one of the selected schools.

Exclusion Criteria:

* Children and their parents who did not give assent and consent to participate in the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Dietary knowledge | 6-months from baseline
  Dietary knowledge will be measured by 24-hour dietary recall questionnaire
  Healthy Eating Index (HEI):
  Scores range from 0 to 100, with higher scores indicating better diet quality. Below 51: Poor diet. 51-80: Needs improvement. Above 80: Good diet
Physical activity education | 6-months from baseline
  Physical activity education will be measured by Global physical activity questionnaire(WHO)
  Total Physical Activity (MET-minutes): The intensity of activities is expressed in Metabolic Equivalent of Task (MET) minutes. MET values are:
  Vigorous-intensity activity: 8.0 METs. Moderate-intensity activity: 4.0 METs. Walking: 4.0 METs. Low Activity: < 600 MET-minutes/week Moderate Activity: 600-2999 MET-minutes/week High Activity: ≥ 3000 MET-minutes/week Sedentary Behavior: More than 8 hours/day of sitting may indicate high sedentary behavior.

SECONDARY OUTCOMES:
Health-related quality of life | 6-months from baseline
  Health-related quality of life will be measured by kids screen questionnaire. 10 items Scoring: Each item is scored on a 5-point Likert scale, summed and transformed into T-scores. Higher scores indicate better overall quality of life.
  T-scores below 40 typically indicate lower quality of life and potential areas of concern.
  T-scores between 40 and 60 are considered within the average range. T-scores above 60 indicate higher than average quality of life.
Body mass index (BMI) | 6-months from baseline
  Body mass index (BMI) will be measured by BMI calculator

CONTACTS AND LOCATIONS:
Locations (1):
- City School Nawab shah, Nawabshah, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The study protocol, statistical plan, and results will be disseminated by publications

REFERENCES:
- [Result] World Health Organisation. (2020, October 19). Noncommunicable diseases: Childhood Overweight and Obesity. Www.who.int. https://www.who.int/news-room/questions-and-answers/item/noncommunicable-diseases-childhood-overweight-and-obesity.
- [Result] Guidelines on Physical Activity, Sedentary Behaviour and Sleep for Children under 5 Years of Age. Geneva: World Health Organization; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK541170/ PMID 31091057
- [Result] Homs C, Berruezo P, Segun G, Estrada L, de Bont J, Riera-Romani J, Carrillo-Alvarez E, Schroder H, Mila R, Gomez SF. Family-based intervention to prevent childhood obesity among school-age children of low socioeconomic status: study protocol of the FIVALIN project. BMC Pediatr. 2021 May 21;21(1):246. doi: 10.1186/s12887-021-02697-x. PMID 34020614
- [Result] Battaglia G, Giustino V, Tabacchi G, Alesi M, Galassi C, Modica C, Palma A, Bellafiore M. Effectiveness of a Physical Education Program on the Motor and Pre-literacy Skills of Preschoolers From the Training-To-Health Project: A Focus on Weight Status. Front Sports Act Living. 2020 Dec 16;2:579421. doi: 10.3389/fspor.2020.579421. eCollection 2020. PMID 33367276
- [Result] L'hôte, E., Hawkins, N., Lead, U., Strategist, S., Levay, K., & Fellow, R. (2021). Prepared for Impact on Urban Health Changing the Childhood Obesity Conversation to Improve Children's Health. https://www.frameworksinstitute.org/wp-content/uploads/2021/04/GSTC-Childhood-obesity-report-032021.pdf
- [Result] Yuksel HS, Sahin FN, Maksimovic N, Drid P, Bianco A. School-Based Intervention Programs for Preventing Obesity and Promoting Physical Activity and Fitness: A Systematic Review. Int J Environ Res Public Health. 2020 Jan 3;17(1):347. doi: 10.3390/ijerph17010347. PMID 31947891